CLINICAL TRIAL: NCT01154621
Title: A Phase I, Double-blind, Randomized, Placebo-Controlled Study to Assess the Safety and Tolerability, and Pharmacokinetics of a Single Dose of AZD9742 in Healthy Elderly Male and Female Volunteers
Brief Title: Assessing the Safety and Tolerability of a Single IV Dose of AZD9742 in Healthy Elderly Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2690C00007
Record Dates: First submitted 2010-06-28; First posted 2010-07-01 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Tolerability; Healthy; Elderly
Keywords: Phase I; Double-blind; Randomized; Placebo-controlled study; Safety and tolerability of single intravenous dose of AZD9742 in healthy elderly volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Single dose of 750mg of intravenous AZD9742 in healthy elderly volunteers
  Interventions: Drug: AZD9742
- 2 (Placebo Comparator): Sterile 5% dextrose solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9742 — Sterile solution, 620 mg (20 mg/mL) in 50 mL vial with a fill volume of 31 mL
  Arms: 1
Drug: Placebo — Sterile 5% dextrose solution
  Arms: 2

SUMMARY:
The aim of this study is to examine the safety and tolerability of a single dose of AZD9742 in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers at age of 65 years or older with suitable veins for cannulation or repeated venipuncture, in good health (based on medical history and physical examination and clinical laboratory tests) as judged by the investigator.
* Female volunteers must be postmenopausal (cessation of regular menses for 12 months and a follicle stimulating hormone level of more than 40IU/L abd estradiol of less than 20ng/mL.
* Male volunteers should be willing to use barrier contraception, ie, condoms, from the day of dosing until 3 months after dosing with the investigational product.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs as judged by Investigator.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of a single intravenous dose of AZD9742 in healthy elderly adults. | The screening period is up to 28 days. Residential period will be a total of 5 days. Follow up will occur between 5 and 10 days after discharge.
  Adverse events, vital signs, electrocardiograms, telemetry, physical exams, and clinical laboratory assessments will be assessed prior to, during, and after treatment

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of a single intravenous dose of AZD9742 in healthy elderly volunteers | Blood and urine samples will be collected for the 4 days while in residence.

CONTACTS AND LOCATIONS:
Overall Officials: Billings W Billings, MD, Principal Investigator — Bio-Kinetic 1816 W. Mt Vernon, Springfield, MO 65802; Colleen Jensen, Study Director — AstraZeneca; Brendan Smyth, Study Chair — AstraZeneca
Locations (1):
- Research Site, Springfield, Missouri, United States